CLINICAL TRIAL: NCT02726269
Title: Helicobacter Pylori Eradication in Mexico With a Levofloxacin-containing Scheme Versus Clarithromycin-based Triple Therapy: a Randomized, Open-label, Non-inferiority, Phase 3b Trial.
Brief Title: Triple Therapy Versus Levofloxacin-based Therapy for Helicobacter Pylori Eradication in Mexico.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asofarma de México S.A de C.V. (Industry)
Collaborators: Hospital Ángeles, Clínica Londres, Mexico City (Unknown); Centro InmunoQ, Mexico City (Unknown); Torre Mayo, Metepec, State of Mexico (Unknown); Hospital Ángeles Metropolitano, Mexico City (Unknown); Centro Médico ABC Observatorio, Mexico City (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASO HO 01
Record Dates: First submitted 2016-03-28; First posted 2016-04-01 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Helicobacter Pylori Gastritis
Keywords: Helicobacter Pylory infections; Levofloxacin; Antibiotic resistance; Clarithromycin; Mutations; Fluorescence; Hybridization
MeSH Terms: interventions — Ofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLA (Clarithro+Lanso+Amoxi) (Active Comparator): Clarithromycin 500 mg bid, Lansoprazole 30 mg bid and Amoxicillin 500 bid, tablets of oral administration, during 10 days.
  Interventions: Drug: CLA (Clarithro+Lanso+Amoxi)
- PLA (Panto+Levoflox+Azithro) (Experimental): Pantoprazole 80 mg od, Levofloxacin 500 mg od and Azithromycin 500 mg od, tablets of oral administration, during 10 days.
  Interventions: Drug: PLA (Panto+Levoflox+Azithro)

INTERVENTIONS:
Drug: CLA (Clarithro+Lanso+Amoxi) — Tablets of oral administration administered to subjects randomized to this group twice daily for 10 days.
  Other Names: Pylopac®, Medix, Mexico
  Arms: CLA (Clarithro+Lanso+Amoxi)
Drug: PLA (Panto+Levoflox+Azithro) — Tablets of oral administration to subjects randomized to this group once daily for 10 days.
  Other Names: Zoltum®, Truxa® (MTV SA, Argentina), Levofloxacino, AsoMex
  Arms: PLA (Panto+Levoflox+Azithro)

SUMMARY:
The goal of this trial is to compare the non-inferiority efficacy and safety of two different treatment schemes: pantoprazole 80 mg + levofloxacin 500 mg + azithromycin 500 mg once daily (PLA, test) vs. clarithromycin 500 mg + lansoprazole 30 mg + amoxicillin 1 g twice daily (CLA, reference), each during 10 days, over Helicobacter Pylori (HP) eradication. Both schemes will be tested in treatment-naive patients, with biopsy-based diagnosis for HP infection. One month after finishing each treatment, C13-urea breath testing will be required to verify HP eradication. Biopsies will also be taken to identify Clarithromycin-resistance mutations in HP strains by fluorescence in situ hybridization (FISH).

DETAILED DESCRIPTION:
This phase IIIb study is a prospective, open-label, randomized, parallel-group, non-inferiority efficacy and safety trial. It will be carried out at four outpatient clinics in two cities placed in Mexico (Mexico City and the town of Toluca). The study was approved by a central Ethics Committee and by COFEPRIS (Mexican Federal Commission for Sanitary Risks Protection) and will be conducted in accordance with Helsinki Declaration for the protection of human subjects and with Good Clinical Practice guidelines.

Two hundred and thirty subjects aged 18 to 65 years, with HP infection proven by endoscopic biopsy and treatment-naïve will be included in the study after signing the informed consent. They will be randomly allocated into one of two groups: Group 1 will receive clarithromycin 500 mg twice daily (bid), amoxicillin 1 g bid, and lansoprazole 30 mg bid (Pylopac®, Medix SA de CV, Mexico); Group 2 will receive azithromycin 500 mg once daily (od) (Truxa®, Laboratorios Monte Verde SA, Argentina), levofloxacin 500 mg od (Laboratorios Asofarma de México SA de CV, Mexico), and pantoprazole 80 mg od (Zoltum®, Laboratorio Monte Verde SA, Argentina). Both groups will receive the treatment for 10 days. Antibiotics will be prescribed after meals, whereas the proton-pump inhibitor will be taken in a fasting condition. No other medication will be allowed until the end of the treatment.

Subjects will be evaluated using the 13C-urea breath test (13C-UBT) four weeks after HP eradication treatment. Eradication of H. pylori will be defined as a negative 13C-UBT. No further medication will be allowed during the four weeks preceding the 13C-UBT.

Regarding safety assessment, blood samples will be collected in a central laboratory following signature of the informed consent and before treatment beginning. An additional blood sample will be drawn at the end of treatment of each group for comparison with initial results. Patient compliance and treatment-related AEs will be assessed at the end of the treatment (except whether the AE is serious, in which case it will be reported immediately and appropriate actions will be decided at that time).

All biopsies will be reviewed by a central pathologist. Endoscopic biopsies will be immediately fixed in 10% buffer formalin, embedded in paraffin, sectioned (4 mm slice thickness), and dehydrated in a series of increasing ethanol/xylol concentration. Each section will be stained with hematoxylin and eosin (H&E). The diagnosis of gastritis will be established in accordance with the updated Sydney system10. Fluorescent in situ hybridization (FISH) will be performed in all biopsies. Briefly, formalin-fixed paraffin-embedded 4-mm tissue sections will be spotted onto slides coated with poly-L-lysine and processed by hexane and ethanol. Hybridization will be done using the commercially available BACTfish H pylori combi kit (Izinta Trading Co. Ltd., Hungary). The probe for H. pylori identification (Hpy 1) (5'CACACCTGACTGACTATCCCG-3') will be labeled with fluorescein isothiocyanate (FITC) that provides a green signal, and the probes that detect the three most prevalent clarithromycin-resistance mutations (ClaR1 (A2143G) 5'CGGGGTCTTCCCGTCTt-3', ClaR2 (A2144G) 5'CGGGGCTCTCCGTCTT-3', and ClaR3 (A21443C) 5-CGGGGTCTTGCCGTCTT-3') will be labeled with red fluorochrome (Cy3). Following hybridization for 90 minutes at 46 °C, sections will be washed with wash buffer twice at 46 °C for 15 minutes. Air-dried sections will be stained with 4', 6' diamino-2-phenylindole (DAPI). Slides will be evaluated using fluorescence Nikon Eclipse 80i microscope. Pictures will be taken with a Nikon DS-Fi1 camera and processed with NIS-Elements 2.1 software.

Continuous variables will be described using means and standard deviation. Efficacy analysis will be based on H. pylori eradication rate in subjects that finished treatment as per protocol. Considering a non-inferiority approach, Group 2 will be considered not inferior to Group 1 if the upper limit of the 95% confidence interval (CI) for the difference in the eradication rate between both groups is lower than the pre-established non-inferiority margin δ = 0.12%. Such margin was selected in accordance with previously published trials performed with the reference combination.

Chi-square test and Student's t-test will be used to compare both groups regarding baseline data, eradication rate, adverse events and biochemical results for safety analysis. P value < 0.05 will be considered significant. IBM SPSS 21 will be used to perform the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult subjects who wish to participate after signing the informed consent.
2. Aged between 18 and 65 years.
3. HP infection diagnosed by endoscopic gastric biopsy.
4. Subjects who fulfill the following HP eradication criteria according to Maastricht 3 Consensus Report:

   * Non ulcer dyspepsia with gastric biopsy positive for HP infection,
   * Uncomplicated duodenal ulcer (without active bleeding, perforation or stenosis) with gastric biopsy positive for HP infection,
   * Uncomplicated benign gastric ulcer (without active bleeding, perforation or stenosis) with gastric biopsy positive for HP infection,
   * Chronic intake of NSAIDs with gastric biopsy positive for HP infection without active gastrointestinal bleeding.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects who have previously received the PLA or CLA treatment.
3. Subjects who are diagnosed by endoscopy with upper gastrointestinal bleeding secondary to active peptic ulcer (gastric or duodenal) with injuries classified in any of the following stages of the Forrest Classification: I-a (Spurting hemorrhage), I-b (Oozing hemorrhage), II-a (Visible vessel) or II-b (Adherent clot).
4. Subjects who are diagnosed by endoscopy with upper gastrointestinal bleeding by erosive gastritis secondary to active NSAID with positive biopsy for HP infection and whose clinical conditions require hospitalization and / or blood transfusion.
5. Subjects with psychiatric disorders including eating disorders.
6. Subjects with chronic degenerative diseases including uncontrolled hepatic, renal or endocrine diseases (except diabetes controlled by oral hypoglycemic agents or controlled hypothyroidism), malabsorption or chronic diarrhea, history of seizures or epilepsy, gastric surgery or subjects with oncological diseases.
7. Subjects with previous allergic reactions to any of the treatment components: Pantoprazole, Amoxicillin, Clarithromycin, Azithromycin or Levofloxacin.
8. Subjects with a history of photosensitivity or tendinitis secondary to quinolones intake.
9. Subjects who are taking any of the following medications:

   * NSAIDS: Fenbufen
   * ergot
   * Oral anticoagulants
   * Cyclosporine
   * Digoxin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
HP eradication rate calculated from negative 13C-urea breath tests. | Four weeks after the end of the allocated treatment.

SECONDARY OUTCOMES:
Determine the frequency of Clarithromycin-resistance mutations by fluorescence in situ hybridization (FISH). | Within a month after taking gastric endoscopy biopsy to confirm the diagnosis of HP infection.
Compare the proportion of Clarithromycin-resistance mutations determined by FISH with the HP eradication rate calculated. | A week after both proportions are calculated.

OTHER OUTCOMES:
Percentage and type of Adverse Events (AEs) and Serious Adverse Events (SAEs) in each group (PLA vs CLA). | Up to a month after the end of both treatments.
Proportion of treatments prematurely suspended due to AEs or SAEs in each group (PLA vs CLA). | Within ten days after each treatment is randomly allocated.

CONTACTS AND LOCATIONS:
Overall Officials: Alma L Ladrón de Guevara, MD, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuadrado-Lavin A, Salcines-Caviedes JR, Carrascosa MF, Dierssen-Sotos T, Cobo M, Campos MR, Ayestaran B, Fernandez-Pousa A, Gonzalez-Colominas E, Aresti-Zarate S, Hernandez M, Pascual EL. Levofloxacin versus clarithromycin in a 10 day triple therapy regimen for first-line Helicobacter pylori eradication: a single-blind randomized clinical trial. J Antimicrob Chemother. 2012 Sep;67(9):2254-9. doi: 10.1093/jac/dks209. Epub 2012 Jun 11. PMID 22687889
- [Background] Chihu L, Ayala G, Mohar A, Hernandez A, Herrera-Goepfert R, Fierros G, Gonzalez-Marquez H, Silva J. Antimicrobial resistance and characterization of Helicobacter pylori strains isolated from Mexican adults with clinical outcome. J Chemother. 2005 Jun;17(3):270-6. doi: 10.1179/joc.2005.17.3.270. PMID 16038520
- [Background] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Derived] Ladron-de-Guevara L, Bornstein-Quevedo L, Gonzalez-Huezo S, Castaneda-Romero B, Costa FG, di Silvio-Lopez M. Helicobacter pylori eradication in Mexico with a levofloxacin-based scheme versus standard triple therapy: Results from an open-label, randomized, noninferiority phase iiib trial. Rev Gastroenterol Mex (Engl Ed). 2019 Jul-Sep;84(3):274-283. doi: 10.1016/j.rgmx.2018.04.005. Epub 2018 Jul 27. English, Spanish. PMID 30060902